CLINICAL TRIAL: NCT00593502
Title: A Double-Blind, Randomized, Placebo-Controlled Study of Early Oseltamivir Treatment of Influenza in Children 1-3 Years of Age
Brief Title: Early Oseltamivir Treatment of Influenza in Children 1-3 Years of Age
Acronym: ETOPOM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital District of Southwestern Finland (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Terho Heikkinen/Consulting Pediatrician, Assistant Professor, Turku University Hospital, Turku, Finland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MV21118; EudraCT 2007-004734-17
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2009-06

CONDITIONS: Influenza
Keywords: influenza; children; acute otitis media; oseltamivir
MeSH Terms: conditions — Influenza, Human; Otitis Media | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Oseltamivir
  Interventions: Drug: oseltamivir
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: oseltamivir — Body weight: ≤ 15 kg, 30 mg twice daily; 15 - ≤ 23 kg, 45 mg twice daily; 23 - ≤ 40 kg, 60 mg twice daily; > 40 kg, 75 mg twice daily, for 5 days
  Other Names: Tamiflu
  Arms: 1
Drug: placebo — The dosage of placebo will be similar to the active drug
  Arms: 2

SUMMARY:
The main purpose of this study is to assess the efficacy of early oseltamivir treatment (started within 24 hours of the onset of influenza symptoms) in preventing the development of acute otitis media as a complication of influenza in children aged 1-3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-3 years
* Fever = or > 38.0 C and at least one respiratory symptom OR fever = or > 38.0 C and a positive influenza rapid test

Exclusion Criteria:

* Confirmed infection with any other respiratory virus than influenza.
* Suspicion of invasive bacterial infection requiring immediate admission to hospital
* Evidence of a poorly controlled underlying medical condition
* Known immunosuppression (malignancy, transplant, drugs)
* Known allergy to oseltamivir or paracetamol
* Received oseltamivir within 4 weeks
* Participation in another clinical trial with an investigational drug

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 409 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Percentage of influenza-infected children in whom acute otitis media develops after the start of study medication | 1-8 days

SECONDARY OUTCOMES:
Time to resolution of fever and other clinical symptoms | 1-21 days

CONTACTS AND LOCATIONS:
Overall Officials: Terho J Heikkinen, MD, Principal Investigator — Turku University Hospital, Turku, Finland
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Background] Heikkinen T, Silvennoinen H, Peltola V, Ziegler T, Vainionpaa R, Vuorinen T, Kainulainen L, Puhakka T, Jartti T, Toikka P, Lehtinen P, Routi T, Juven T. Burden of influenza in children in the community. J Infect Dis. 2004 Oct 15;190(8):1369-73. doi: 10.1086/424527. Epub 2004 Sep 15. PMID 15378427
- [Background] Whitley RJ, Hayden FG, Reisinger KS, Young N, Dutkowski R, Ipe D, Mills RG, Ward P. Oral oseltamivir treatment of influenza in children. Pediatr Infect Dis J. 2001 Feb;20(2):127-33. doi: 10.1097/00006454-200102000-00002. PMID 11224828
- [Derived] Heinonen S, Silvennoinen H, Lehtinen P, Vainionpaa R, Ziegler T, Heikkinen T. Effectiveness of inactivated influenza vaccine in children aged 9 months to 3 years: an observational cohort study. Lancet Infect Dis. 2011 Jan;11(1):23-9. doi: 10.1016/S1473-3099(10)70255-3. Epub 2010 Nov 22. PMID 21106443
- [Derived] Heinonen S, Silvennoinen H, Lehtinen P, Vainionpaa R, Vahlberg T, Ziegler T, Ikonen N, Puhakka T, Heikkinen T. Early oseltamivir treatment of influenza in children 1-3 years of age: a randomized controlled trial. Clin Infect Dis. 2010 Oct 15;51(8):887-94. doi: 10.1086/656408. PMID 20815736